CLINICAL TRIAL: NCT04349891
Title: Transcutaneous Electroacupuncture for Gastrointestinal Motility Disorders
Acronym: TEA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left Johns Hopkins University
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00247402
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEA at ST36 and PC6 first and then sham TEA (Experimental): Patients in this group will be treated with TEA at ST36 and PC6 for 4 weeks, followed with a 2-week washout period and another 4-week period with sham TEA.
  Interventions: Device: Transcutaneous Electroacupuncture; Device: Sham TEA
- Sham-TEA and then TEA ST36 and PC6 (Experimental): Patients in this group will be treated with sham-TEA for 4 weeks, followed with a 2-week washout period and another 4-week period with TEA at ST36 and PC6.
  Interventions: Device: Transcutaneous Electroacupuncture; Device: Sham TEA

INTERVENTIONS:
Device: Transcutaneous Electroacupuncture — Weak electrical current will be generated by the device and delivered via skin surface electrodes to acupuncture points related to gastrointestinal functions.
Device: Sham TEA — Sham will be delivered via skin surface electrodes to acupuncture points related to gastrointestinal functions.

SUMMARY:
Gastrointestinal (GI) dysmotility is common in GI motility disorders, such as functional dyspepsia (FD) gastroparesis and chronic constipation. The symptoms of GI dysmotility include abdominal discomfort or pain, early satiety, nausea, vomiting, abdominal distension, bloating, anorexia and reduced bowel movement. . Medical treatment for GI motility disorders is very limited in the US. Acupuncture has frequently been used for treatment of GI ailments in Eastern countries. The most commonly used acupuncture points (acupoints) for focused treatment of GI symptoms are the Neiguan (PC6) and the Zusanli (ST36) points. Electroacupuncture (EA) at PC6 and ST36 has been reported to accelerate gastrointestinal motility in both animals and human.

Recently, the investigators have studied the feasibility of transcutaneous electroacupuncture (TEA): electrical stimulation is applied to acupoints via surface electrodes without needles, similar to the commercial available transcutaneous electrical nerve stimulation (TENS) but applied to acupoints. The investigators hypothesize that TEA as a new treatment option, improves GI symptoms in patients with FD, gastroparesis or constipation, improves GI motility and therefore improves quality of life of the patients.

The success of this project will lead to a noninvasive and convenient therapy for treating GI motility disorders. The proposed TEA method is expected to improve gastric and colonic functions and thus improve quality of life. In addition, the proposed TEA method and device are self-administrative after training during the first office visit. It provides a long-term treatment option for both FD, gastroparesis and chronic constipation.

ELIGIBILITY:
Inclusion criteria for FD patients

* Bothersome postprandial fullness
* Symptoms of early satiation, epigastric pain, epigastric burning during the last 3 months
* No evidence of structural disease including at upper endoscopy that is likely to explain the symptoms.
* Males and females between ages 18-80 yrs;
* Subjects with high probability for compliance and completion of the study.

Inclusion criteria for chronic constipation patients

* Satisfying Rome IV criteria for diagnosis of functional constipation;
* abdominal X-ray or anorectal manometry test during the past 3 months indicating delayed colonic transit (more than 20% ingested markers are retained) or abnormal colonic motility;
* ages 18-80 years;
* no constipation medication for a minimum of 1 week before enrollment except for rescue agents (stimulant laxatives, such as bisacodyl);
* willing to comply with the treatment regimen.

Inclusion criteria for gastroparesis patients

* At least one severe gastroparetic symptom or two moderate gastroparetic symptoms (see assessment of gastroparetic symptoms);
* Abnormal gastric emptying diagnosed during the past year;
* Males and females between ages 18-80 yrs;
* Subjects with high probability for compliance and completion of the study.
* Upper endoscopy or upper GI within last 2 years showing no evidence of gastric bezoar, stricture, or peptic ulcer.

Exclusion criteria:

* History of gastric bezoar or diverticulitis.
* Severe daily abdominal pain requiring narcotic medications.
* Previous gastro-esophageal surgery including vagotomy, fundoplication, gastric bypass, ulcer surgery.
* Prior GI surgery except for uncomplicated appendectomy and laparoscopic cholecystectomy;
* Surgery within the past 3 months.
* Female of childbearing age who is not practicing birth control and/or is pregnant or lactating. (Confirm with urine pregnancy test).
* Those who have been treated with acupuncture or those who are familiar with acupuncture points.
* Anyone with an implantable cardiac pacemaker or defibrillator.
* unable to give informed consent;
* taking prokinetics, anticholinergic or dopaminergic agents;
* history of gastrointestinal surgery;
* pregnant or preparing to conceive a child;
* diabetes;
* allergic to skin preparation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Pasricha, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Once the inclusion and exclusion criteria were satisfied, patients were assigned randomly to either the treatment group or the sham group. No subjects were excluded prior to the assignment of participants to their respective groups.
Period: First Intervention - 4 Weeks
Arm/Group | TEA at ST36 and PC6 First and Then Sham TEA | Sham-TEA and Then TEA ST36 and PC6
Started | 15 | 12
Completed | 11 | 7
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Adverse Event | 1 | 1
Period: Washout - 2 Weeks
Arm/Group | TEA at ST36 and PC6 First and Then Sham TEA | Sham-TEA and Then TEA ST36 and PC6
Started | 11 | 7
Completed | 10 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention - 4 Weeks
Arm/Group | TEA at ST36 and PC6 First and Then Sham TEA | Sham-TEA and Then TEA ST36 and PC6
Started | 10 | 7
Completed | 8 | 7
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TEA at ST36 and PC6 First and Then Sham TEA | Sham-TEA and Then TEA ST36 and PC6 | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 10 | 25
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (7.5) | 40.9 (2) | 37.2 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 12 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 12 | 27
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.34 (5.7) | 22.01 (4.8) | 22.8 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Gastroparesis Cardinal Symptom Index (GCSI) Score
Description: The effect of TEA on gastrointestinal dysmotility syndrome by changes in the score of the Gastroparesis Cardinal Symptom Index (GCSI) including 9 symptoms: nausea (feeling sick to your stomach as if you were going to vomit or throw up), retching (heaving as if to vomit, but nothing comes up), vomiting, stomach fullness, not able to finish a normal sized meal, feeling excessively full after meals, loss of appetite, bloating (feeling like you need to loose your clothes) and stomach or belly visibly larger. Each symptom will be graded from 0 to 5 (none, very mild, mild, moderate, severe and very severe). GCSI total score can range from 0 to 5, with higher scores reflecting greater symptom severity. The
Time Frame: Up to 10 weeks
Population: The number of participants analyzed are the ones who completed each study intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TEA at ST36 and PC6 First and Then Sham TEA | Sham-TEA and Then TEA ST36 and PC6
Number analyzed (Participants) | 11 | 7
score on a scale
  First Intervention | 2.60 (0.88) | 2.84 (1.21)
  Washout: number analyzed (Participants) | 10 | 7
  Washout | 2.58 (0.81) | 2.74 (1.21)
  Second intervention: number analyzed (Participants) | 8 | 7
  Second intervention | 2.22 (0.58) | 2.84 (1.14)

2. Secondary Outcome: Change in Number of Spontaneous Complete Bowel Movements
Description: The effect of TEA on gastrointestinal dysmotility syndrome by changes in the number of Spontaneous Complete Bowel Movements.
Time Frame: Up to 10 weeks
Population: Patients who provided data at the end of each study intervention.
Measure: Mean (Standard Deviation); unit: number of bowel movements
Arm/Group | TEA at ST36 and PC6 First and Then Sham TEA | Sham-TEA and Then TEA ST36 and PC6
Number analyzed (Participants) | 11 | 7
number of bowel movements
  First intervention - end of the 4th week of study participation. | 8.79 (13.74) | 11.45 (17.02)
  Washout - end of 6th week: number analyzed (Participants) | 10 | 7
  Washout - end of 6th week | 12.88 (22.84) | 11.07 (12.93)
  Second intervention - end of the 10th week.: number analyzed (Participants) | 8 | 7
  Second intervention - end of the 10th week. | 9.38 (10.46) | 10.68 (11.76)

3. Secondary Outcome: Change in the Patient Assessment of Constipation (PAC-SYN) Score
Description: The effect of TEA on gastrointestinal dysmotility syndrome by changes in the score of Patient Assessment of Constipation (PAC-SYN). This questionnaire asks about constipation in the past 2 weeks. Symptoms include: abdominal discomfort, abdominal pain, bloating, stomach cramps, painful bowel movements, rectal burning, rectal bleeding, incomplete bowel movement, hardness of stool, size of bowel movements, straining and feeling to pass a bowel without success. Each symptom will be scored between 1 to 4 being 1 for mild symptoms; 2 for moderate; 3 for severe and 4 for very severe. A total PAC-SYM score ranges from 0 to 48 with a low score indicating fewer symptoms and of lower severity.
Time Frame: Up to 10 weeks
Population: Patients who provided data at the end of each study intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TEA at ST36 and PC6 First and Then Sham TEA | Sham-TEA and Then TEA ST36 and PC6
Number analyzed (Participants) | 11 | 7
score on a scale
  First Intervention - End of the 4th week | 17.14 (8.31) | 17.30 (10.74)
  Washout - End of 6th week: number analyzed (Participants) | 10 | 7
  Washout - End of 6th week | 16.83 (9.64) | 16.21 (11.12)
  Second Intervention - End of 10th week: number analyzed (Participants) | 8 | 7
  Second Intervention - End of 10th week | 13.9 (8.47) | 17.03 (10.68)

4. Secondary Outcome: Change in Quality of Life as Assessed by the Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life Scale
Description: The effect of TEA on quality of life assessed by the Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life (PAGI-QoL). The PAGI-QoL instrument consists of 30 items, each with response options based on a 6-point scale and with a recall period of the previous 2 weeks. The items are grouped into 5 dimensions: Daily Activities, Clothing, Diet and Food Habits, Relationship and Psychological Well-being and Distress. A score per dimension as well as a total score can be calculated. The PAGI-QOL scores range from 0 (lowest QoL) to 5 (highest QoL). There is not an established PAC-QOL score for the diagnosis of constipation.
Time Frame: Up to 10 weeks
Population: Patients who provided data at the end of each study intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TEA at ST36 and PC6 First and Then Sham TEA | Sham-TEA and Then TEA ST36 and PC6
Number analyzed (Participants) | 11 | 7
score on a scale
  First intervention - End of 4th week. | 1.76 (0.64) | 1.40 (0.50)
  Washout - End of 6th week.: number analyzed (Participants) | 10 | 7
  Washout - End of 6th week. | 1.86 (0.62) | 1.42 (0.53)
  Second intervention - End of the 10th week.: number analyzed (Participants) | 8 | 7
  Second intervention - End of the 10th week. | 1.72 (0.56) | 1.41 (0.50)

5. Secondary Outcome: Change in Dimensions of Health as Assessed by the Short Form (SF-36v2) Health Survey
Description: The effect of TEA on quality of life assessed by the SF-36v2 Health Survey. The SF-36v2 is a 36-item, self-report measure designed to assess quality of life in patients. This measure also provides two summary scores (physical and mental health) and eight scale scores. The eight sections are: vitality, physical functioning, bodily pain and general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability, i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The subscales will be combined to report average mean score.
Time Frame: Up to 10 weeks
Population: Patients who provided data at the end of each study intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TEA at ST36 and PC6 First and Then Sham TEA | Sham-TEA and Then TEA ST36 and PC6
Number analyzed (Participants) | 15 | 12
score on a scale
  First Intervention - End of 4th Week: number analyzed (Participants) | 11 | 7
  First Intervention - End of 4th Week | 45.83 (9.63) | 51.21 (9.70)
  Wash out - End of 6th week.: number analyzed (Participants) | 10 | 7
  Wash out - End of 6th week. | 43.21 (8.66) | 50.95 (8.74)
  Second intervention - End of 10th week: number analyzed (Participants) | 8 | 7
  Second intervention - End of 10th week | 44.47 (11.45) | 54.17 (7.72)

ADVERSE EVENTS:
Time Frame: Up to 10 weeks
Description: Serious Adverse Events and All-cause mortality were not collected.
Groups:
- TEA at ST36 and PC6: Patients in this group received TEA at ST36 and PC6 for 4 weeks
- Sham - TEA: Patients in this group received sham-TEA for 4 weeks
Arm/Group | TEA at ST36 and PC6 | Sham - TEA
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/22 | 1/22
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TEA at ST36 and PC6 (N=22) | Sham - TEA (N=22)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT04349891/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT04349891/ICF_001.pdf